CLINICAL TRIAL: NCT00514683
Title: A 12 Month, Double Blind, Randomized, Placebo-controlled Trial Evaluating the Effect of BIBF 1120 Administered at Oral Doses of 50 mg qd, 50 mg Bid, 100 mg Bid and 150 mg Bid on Forced Vital Capacity Decline During One Year, in Patients With Idiopathic Pulmonary Fibrosis, With Optional Active Treatment Extension Until Last Patient Out.
Brief Title: Safety And Efficacy of BIBF 1120 in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.30
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

ARMS (5):
- dose 1 (Experimental): low dose BIBF1120 once daily
  Interventions: Drug: low dose BIBF1120 once daily
- dose 2 (Experimental): low dose BIBF 1120 twice daily
  Interventions: Drug: low dose BIBF 1120 twice daily
- dose 3 (Experimental): intermediate dose BIBF 1120 twice daily
  Interventions: Drug: intermediate dose BIBF 1120 twice daily
- dose 4 (Experimental): high dose BIBF 1120 twice daily
  Interventions: Drug: high dose BIBF 1120 twice daily
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: low dose BIBF1120 once daily — low dose BIBF1120 once daily
  Arms: dose 1
Drug: low dose BIBF 1120 twice daily — low dose BIBF 1120 twice daily
  Arms: dose 2
Drug: intermediate dose BIBF 1120 twice daily — intermediate dose BIBF 1120 twice daily
  Arms: dose 3
Drug: high dose BIBF 1120 twice daily — high dose BIBF 1120 twice daily
  Arms: dose 4
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The general purpose of this trial is to investigate the efficacy and safety of 4 dose strategies of BIBF 1120 treatment for 12 months, compared to placebo in patients with idiopathic pulmonary fibrosis.

The primary objective of this study is to demonstrate whether at least one dose strategy is superior to placebo in patients with IPF, in modifying the rate of decline of Forced Vital Capacity (FVC).

As a secondary objective, additional parameters will be assessed in order to differentiate between dose strategies on the basis of safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Patient >40 years
2. Written informed consent signed prior to entry into the study
3. IPF diagnosed (according to ATS / ERS criteria) less than 5 years prior to screening visit.
4. HRCT within 12 months of randomisation and biopsy (the latter if needed to fulfil ATS/ERS criteria) centrally reviewed and consistent with diagnosis.
5. FVC>50 % of predicted value

   Predicted normal values will be calculated according to ESCS (R94-1408):

   Males :

   FVC predicted (L) = 5.76 x height (meters)- 0.026 x age (years) -4.34

   Females :

   FVC predicted (L) = 4.43 x height (meters)- 0.026 x age (years) -2.89
6. Single breath DLCO (corrected for Hb) 30 - 79% inclusive of predicted .

   Different sites may use different prediction formulas, based on the method used to measure DLco. In any case, the method used must be in compliance with the ATS/ERS guideline on DLCO measurements (R06-2002), and the prediction formula appropriate for that method. Raw data (gas mixture, equation used for prediction of normal, further adjustments made if so) must be traced.

   Adjustment for haemoglobin (R06-2002):

   Males :

   DLCO predicted for Hb = DLCO predicted x (1.7Hb/[10.22+Hb])

   Females :

   DLCO predicted for Hb = DLCO predicted x (1.7Hb/[9.38+Hb]) where Hb is expressed in g/dL-1
7. PaO2 >= 55 mmHg (sea level to 1500 m) or 50 mmHg (above 1500 m) room air

Exclusion Criteria:

1. AST, ALT > 1.5 x ULN ;
2. Bilirubin > 1.5 x ULN
3. Relevant airways obstruction
4. Continuous oxygen supplementation at randomisation (defined as > 15 hours supplemental oxygen per day).
5. Active infection at screening or randomisation.
6. Neutrophils < 1500 / mm3
7. International normalised ratio (INR) > 1.5 and/or Partial thromboplastin time (PTT) > 1.5 x ULN ;
8. Platelets < 100 000 /mL
9. Haemoglobin < 9.0 g/dL
10. In the opinion of the Investigator, patient is likely to have lung transplantation during study
11. Life expectancy for disease other than IPF < 2.5 years (Investigator assessment).
12. Other disease that may interfere with testing procedures or in judgement of Investigator may interfere with trial participation or may put the patient at risk when participating to this trial.

    * Myocardial infarction during the previous 6 months
    * Unstable angina during the previous month
13. Other investigational therapy received within 8 weeks prior to screening visit.
14. Pregnant women or women who are breast feeding or of child bearing potential not using a highly effective method of birth control for at least one month prior to enrolment.
15. Sexually active males not committing to using condoms during the course of the study (except if their partner is not of childbearing potential).
16. Known or suspected active alcohol or drug abuse.
17. Bleeding risk : Known inherited predisposition to bleeding, patients who require full-dose anticoagulation, Patients who require full-dose antiplatelet therapy, History of hemorrhagic CNS event within 12 months prior to screening , Any of the following within 3 months prior to screening : Gross / frank haemoptysis or haematuria, Active gastro-intestinal bleeding or ulcers, Major injury or surgery
18. Thrombotic risk
19. Surgical procedures planned to occur during trial period.
20. Coagulopathy
21. Uncontrolled systemic arterial hypertension
22. known hypersensitivity to lactose or any component of the study medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (92):
- 1199.30.54002 Boehringer Ingelheim Investigational Site, Mendoza, Argentina
- Australia (4):
  - 1199.30.61005 Boehringer Ingelheim Investigational Site, South Brisbane, Queensland
  - 1199.30.61003 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1199.30.61004 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 1199.30.61001 Royal Perth Hospital, Perth, Western Australia
- Belgium (3):
  - 1199.30.32004 Boehringer Ingelheim Investigational Site, Brussels
  - 1199.30.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1199.30.32002 Boehringer Ingelheim Investigational Site, Yvoir
- Brazil (2):
  - 1199.30.55002 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1199.30.55001 Boehringer Ingelheim Investigational Site, Vila Clementino
- Bulgaria (2):
  - 1199.30.06004 Boehringer Ingelheim Investigational Site, Sofia
  - 1199.30.06005 Boehringer Ingelheim Investigational Site, Sofia
- Canada (2):
  - 1199.30.01003 Division of Respirology, Halifax, Nova Scotia
  - 1199.30.01002 St. Joseph's Healthcare, Hamilton, Ontario
- 1199.30.56001 Boehringer Ingelheim Investigational Site, Providencia, Chile
- China (5):
  - 1199.30.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1199.30.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1199.30.86005 Boehringer Ingelheim Investigational Site, Nanjing
  - 1199.30.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 1199.30.86004 Boehringer Ingelheim Investigational Site, Shenyang
- Czechia (2):
  - 1199.30.42002 Boehringer Ingelheim Investigational Site, Prague
  - 1199.30.42001 Boehringer Ingelheim Investigational Site, Ústí nad Labem
- France (9):
  - 1199.30.3302A Boehringer Ingelheim Investigational Site, Bobigny
  - 1199.30.3306A Boehringer Ingelheim Investigational Site, Dijon
  - 1199.30.3303A Boehringer Ingelheim Investigational Site, Grenoble
  - 1199.30.3305A Boehringer Ingelheim Investigational Site, Lille
  - 1199.30.3305B Boehringer Ingelheim Investigational Site, Lille
  - 1199.30.3305C Boehringer Ingelheim Investigational Site, Lille
  - 1199.30.3304C Boehringer Ingelheim Investigational Site, Montpellier
  - 1199.30.3307A Boehringer Ingelheim Investigational Site, Nice
  - 1199.30.3301A Boehringer Ingelheim Investigational Site, Paris
- Germany (9):
  - 1199.30.49008 Boehringer Ingelheim Investigational Site, Bad Berka
  - 1199.30.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1199.30.49006 Boehringer Ingelheim Investigational Site, Donaustauf
  - 1199.30.49001 Boehringer Ingelheim Investigational Site, Essen
  - 1199.30.49002 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1199.30.49003 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1199.30.49009 Boehringer Ingelheim Investigational Site, Leipzig
  - 1199.30.49004 Boehringer Ingelheim Investigational Site, Mainz
  - 1199.30.49005 Boehringer Ingelheim Investigational Site, München
- Greece (3):
  - 1199.30.30004 Boehringer Ingelheim Investigational Site, Alexandroupoli
  - 1199.30.30001 Boehringer Ingelheim Investigational Site, Heraklion
  - 1199.30.30002 Boehringer Ingelheim Investigational Site, Larissa
- Hungary (5):
  - 1199.30.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 1199.30.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1199.30.36004 Boehringer Ingelheim Investigational Site, Deszk
  - 1199.30.36001 Boehringer Ingelheim Investigational Site, Pécs
  - 1199.30.36005 Boehringer Ingelheim Investigational Site, Székesfehérvár
- 1199.30.35301 Mater Misericordiae Hospital, Dublin, Ireland
- Italy (10):
  - 1199.30.39008 Boehringer Ingelheim Investigational Site, Ascoli Piceno
  - 1199.30.39013 Boehringer Ingelheim Investigational Site, Busto Arsizio (va)
  - 1199.30.39007 Boehringer Ingelheim Investigational Site, Milan
  - 1199.30.39001 Boehringer Ingelheim Investigational Site, Modena
  - 1199.30.39012 Boehringer Ingelheim Investigational Site, Napoli
  - 1199.30.39009 Boehringer Ingelheim Investigational Site, Pavia
  - 1199.30.39011 Boehringer Ingelheim Investigational Site, Roma
  - 1199.30.39010 Boehringer Ingelheim Investigational Site, Siena
  - 1199.30.39003 Boehringer Ingelheim Investigational Site, Terni
  - 1199.30.39004 Boehringer Ingelheim Investigational Site, Trieste
- 1199.30.52001 Boehringer Ingelheim Investigational Site, Distrito Federal, Mexico
- 1199.30.31002 Boehringer Ingelheim Investigational Site, Nieuwegein, Netherlands
- Portugal (6):
  - 1199.30.35105 Boehringer Ingelheim Investigational Site, Coimbra
  - 1199.30.35106 Boehringer Ingelheim Investigational Site, Coimbra
  - 1199.30.35107 Boehringer Ingelheim Investigational Site, Lisbon
  - 1199.30.35108 Boehringer Ingelheim Investigational Site, Lisbon
  - 1199.30.35109 Boehringer Ingelheim Investigational Site, Lisbon
  - 1199.30.35101 Boehringer Ingelheim Investigational Site, Porto
- Russia (3):
  - 1199.30.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 1199.30.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 1199.30.07003 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (3):
  - 1199.30.27001 Boehringer Ingelheim Investigational Site, Bellville
  - 1199.30.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 1199.30.27002 Boehringer Ingelheim Investigational Site, Tygerberg
- South Korea (5):
  - 1199.30.82002 Boehringer Ingelheim Investigational Site, Gyunggido
  - 1199.30.82004 Boehringer Ingelheim Investigational Site, Incheon
  - 1199.30.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.30.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.30.82005 Boehringer Ingelheim Investigational Site, Seoul
- Spain (2):
  - 1199.30.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1199.30.34002 Boehringer Ingelheim Investigational Site, Valencia
- Taiwan (5):
  - 1199.30.88605 Boehringer Ingelheim Investigational Site, Taichung
  - 1199.30.88601 National Taiwan University, Taipei
  - 1199.30.88603 Tri-service General Hospital, Taipei
  - 1199.30.88606 Boehringer Ingelheim Investigational Site, Taipei
  - 1199.30.88604 Chang Gung Memorial Hosp-Linkou, Taoyuan District
- Turkey (Türkiye) (2):
  - 1199.30.90001 Boehringer Ingelheim Investigational Site, Ankara
  - 1199.30.90002 Boehringer Ingelheim Investigational Site, Istanbul
- United Kingdom (5):
  - 1199.30.44006 Boehringer Ingelheim Investigational Site, Aberdeen
  - 1199.30.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 1199.30.44005 Boehringer Ingelheim Investigational Site, Birmingham
  - 1199.30.44007 Boehringer Ingelheim Investigational Site, Manchester
  - 1199.30.44001 Boehringer Ingelheim Investigational Site, Westbury on Trym

REFERENCES:
- [Derived] Glaspole I, Bonella F, Bargagli E, Glassberg MK, Caro F, Stansen W, Quaresma M, Orsatti L, Bendstrup E. Efficacy and safety of nintedanib in patients with idiopathic pulmonary fibrosis who are elderly or have comorbidities. Respir Res. 2021 Apr 26;22(1):125. doi: 10.1186/s12931-021-01695-y. PMID 33902584
- [Derived] Richeldi L, Kreuter M, Selman M, Crestani B, Kirsten AM, Wuyts WA, Xu Z, Bernois K, Stowasser S, Quaresma M, Costabel U. Long-term treatment of patients with idiopathic pulmonary fibrosis with nintedanib: results from the TOMORROW trial and its open-label extension. Thorax. 2018 Jun;73(6):581-583. doi: 10.1136/thoraxjnl-2016-209701. Epub 2017 Oct 9. PMID 28993537
- [Derived] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260
- [Derived] Richeldi L, Costabel U, Selman M, Kim DS, Hansell DM, Nicholson AG, Brown KK, Flaherty KR, Noble PW, Raghu G, Brun M, Gupta A, Juhel N, Kluglich M, du Bois RM. Efficacy of a tyrosine kinase inhibitor in idiopathic pulmonary fibrosis. N Engl J Med. 2011 Sep 22;365(12):1079-87. doi: 10.1056/NEJMoa1103690. PMID 21992121

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients were treated with matching Placebo.
- Nintedanib 50 qd: Patients were treated with 50mg nintedanib once daily
- Nintedanib 50 Bid: Patients were treated with 50mg nintedanib twice daily
- Nintedanib 100 Bid: Patients were treated with 100mg nintedanib twice daily
- Nintedanib 150 Bid: Patients were treated with 150mg nintedanib twice daily
Period: Overall Study
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Started | 87 (Randomised) | 87 (Randomised) | 86 (Randomised) | 86 (Randomised) | 86 (Randomised)
Completed | 61 | 62 | 68 | 72 | 53
Not Completed | 26 | 25 | 18 | 14 | 33
Not completed — Not treated | 2 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 21 | 20 | 15 | 13 | 27
Not completed — Protocol Violation | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0 | 4
Not completed — Reason other than listed above | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set: This patient set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid | Total
Number analyzed (Participants) | 85 | 86 | 86 | 86 | 85 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.57) | 65.3 (9.42) | 64.9 (8.48) | 65.1 (8.63) | 65.4 (7.82) | 65.1 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 24 | 21 | 20 | 108
  Male | 63 | 65 | 62 | 65 | 65 | 320

OUTCOME MEASURES:

1. Primary Outcome: Rate of Decline in FVC
Description: Rate of decline in Forced Vital Capacity (FVC) evaluated from baseline until 52 weeks of treatment.
  The means presents actually the adjusted rate based on a MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time.
Time Frame: Baseline until 52 weeks
Population: Observed Case (OC): This method was used for the replacement of missing values.
  Randomised set: This patient set includes all randomised patients whether treated or not.
Measure: Mean (Standard Error); unit: Liters/year
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 83 | 85 | 86 | 85 | 84
Liters/year | -0.190 (0.036) | -0.174 (0.037) | -0.210 (0.035) | -0.162 (0.035) | -0.060 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8530, Mixed Models Analysis — The p-value presented is computed in the course of the closing testing procedure; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.086 to 0.118], Standard Error of Mean 0.052 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7558, Mixed Models Analysis — The p-value from the hierarchical testing procedure was calculated as a sensitivity analysis; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.7920, Mixed Models Analysis — The p-value presented is computed in the course of the closing testing procedure; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time; Mean Difference (Final Values) = -0.020, 95% CI 2-sided [-0.119 to 0.080], Standard Error of Mean 0.051 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6991, Mixed Models Analysis — The p-value from the hierarchical testing procedure was calculated as a sensitivity analysis; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time
Statistical Analysis 5: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.8530, Mixed Models Analysis — The p-value presented is computed in the course of the closing testing procedure; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.071 to 0.128], Standard Error of Mean 0.051 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 6: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.5736, Mixed Models Analysis — Additionally the p-value from the hierarchical testing procedure was calculated as a sensitivity analysis; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time
Statistical Analysis 7: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0639, Mixed Models Analysis — The p-value presented is computed in the course of the closing testing procedure; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.027 to 0.235], Standard Error of Mean 0.053 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 8: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis — Additionally the p-value from the hierarchical testing procedure was calculated as a sensitivity analysis; MMRM with fixed terms for treatment*time, gender*height, gender*age and random terms for patient effect, patient*time

2. Secondary Outcome: Absolute Change From Baseline in FVC%Pred
Description: Change from baseline in percentage of predicted Forced Vital Capacity (FVC%pred) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline and region.
Time Frame: Baseline and 52 weeks
Population: Last Observation Carried Forward (LOCF): This method was used for the replacement of missing values.
  Randomised set: This patient set includes all randomised patients whether treated or not.
Measure: Mean (Standard Error); unit: percentage of predicted FVC
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
percentage of predicted FVC | -6.00 (1.019) | -4.58 (1.029) | -4.90 (0.984) | -3.15 (1.004) | -1.04 (0.990)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.2774, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.43, 95% CI 2-sided [-1.15 to 4.01], Standard Error of Mean 1.312 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.4014, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [-1.48 to 3.68], Standard Error of Mean 1.312 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0314, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [0.26 to 5.46], Standard Error of Mean 1.324 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0002, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 4.97, 95% CI 2-sided [2.37 to 7.56], Standard Error of Mean 1.319 — Mean difference to placebo is calculated. Negative change indicates worsening

3. Secondary Outcome: Absolute Change From Baseline in FVC
Description: Change from baseline in percentage of absolute Forced Vital Capacity (FVC) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline and region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
Liters | -0.23 (0.036) | -0.18 (0.036) | -0.19 (0.035) | -0.13 (0.035) | -0.06 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.3644, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.05 to 0.13], Standard Error of Mean 0.046 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.4525, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.06 to 0.13], Standard Error of Mean 0.046 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0471, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.00 to 0.18], Standard Error of Mean 0.046 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.08 to 0.26], Standard Error of Mean 0.046 — Mean difference to placebo is calculated. Negative change indicates worsening

4. Secondary Outcome: Relative Change From Baseline in FVC%Pred
Description: Percent change from baseline in percentage of predicted Forced Vital Capacity (FVC%pred) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline and region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
percentage of change | -7.28 (1.321) | -6.37 (1.334) | -6.42 (1.277) | -3.47 (1.302) | -1.81 (1.283)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.5920, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-2.43 to 4.26], Standard Error of Mean 1.702 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6155, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-2.49 to 4.20], Standard Error of Mean 1.702 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0271, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 3.81, 95% CI 2-sided [0.43 to 7.18], Standard Error of Mean 1.716 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0015, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 5.47, 95% CI 2-sided [2.11 to 8.83], Standard Error of Mean 1.710 — Mean difference to placebo is calculated. Negative change indicates worsening

5. Secondary Outcome: Relative Change From Baseline in FVC
Description: Percent change from baseline in absolute Forced Vital Capacity (FVC) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline and region
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
percentage change | -7.96 (1.314) | -6.98 (1.327) | -7.16 (1.272) | -4.13 (1.285) | -2.52 (1.277)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.5601, ANCOVA — ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [-2.34 to 4.31], Standard Error of Mean 1.692 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6366, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-2.53 to 4.13], Standard Error of Mean 1.694 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0246, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 3.84, 95% CI 2-sided [0.49 to 7.18], Standard Error of Mean 1.702 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0015, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 5.44, 95% CI 2-sided [2.10 to 8.78], Standard Error of Mean 1.700 — Mean difference to placebo is calculated. Negative change indicates worsening

6. Secondary Outcome: Number of Participants With Change From Baseline in FVC by Categories
Description: Change from baseline in percentage of Forced Vital Capacity (FVC) at 52 weeks in below mentioned categories:
  1. Decrease > 10% or 200mL
  2. Change within <= 10% or <=200 mL
  3. Increase > 10% or 200mL
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Number; unit: participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
participants
  Decrease > 10% or 200mL | 37 | 35 | 41 | 30 | 20
  Change within <= 10% or <=200mL | 41 | 44 | 39 | 46 | 52
  Increase > 10% or 200mL | 6 | 6 | 6 | 9 | 12
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7543, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.911, 95% CI 2-sided [0.506 to 1.637] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6704, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.136, 95% CI 2-sided [0.631 to 2.045] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1649, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.657, 95% CI 2-sided [0.363 to 1.189] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0041, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.415, 95% CI 2-sided [0.227 to 0.757] — Odds ratio lower than 1 favours the treatment group over placebo

7. Secondary Outcome: Survival (All Causes of Death and Lung-transplant Free)
Description: Survival (all causes of death and lung-transplant free) at 52 weeks, based on overall mortality and on-treatment survival.
  Failure means participants with event and Censored means participants with no event.
Time Frame: 52 weeks
Population: OC-Randomised set
Measure: Number; unit: participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
participants
  Failure | 9 | 11 | 3 | 4 | 7
  Censored | 78 | 76 | 83 | 82 | 79
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.5882, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 1.278, 95% CI 2-sided [0.526 to 3.102] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.0653, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.290, 95% CI 2-sided [0.078 to 1.081] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0847, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.350, 95% CI 2-sided [0.106 to 1.154] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.5383, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.271 to 1.977] — Hazard ratio lower than 1 favours the treatment group over placebo

8. Secondary Outcome: Absolute Change From Baseline in SpO2 at Rest
Description: Absolute change from baseline in oxygen saturation (SpO2) at rest.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Percentage of SpO2
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 82 | 82 | 86 | 84 | 83
Percentage of SpO2 | -1.29 (0.373) [-2.03 to -0.56] | -0.86 (0.380) [-1.60 to -0.11] | -0.97 (0.357) [-1.67 to -0.27] | 0.06 (0.363) [-0.65 to 0.78] | -0.18 (0.360) [-0.89 to 0.53]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.3658, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.51 to 1.39], Standard Error of Mean 0.483 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.4956, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.61 to 1.27], Standard Error of Mean 0.478 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0051, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [0.41 to 2.31], Standard Error of Mean 0.482 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0211, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.17 to 2.07], Standard Error of Mean 0.483 — Mean difference to placebo is calculated. Negative change indicates worsening

9. Secondary Outcome: Absolute Change From Baseline in SpO2 at Rest by Categories
Description: Absolute change from baseline in oxygen saturation (SpO2) at rest by below mentioned categories:
  SpO2 (non-invasive) at 52 weeks:
  1. Decrease > 4% SpO2
  2. Change within +/- 4% SpO2
  3. Increase > 4% SpO2
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 82 | 82 | 86 | 84 | 83
percentage of participants
  Decrease > 4% | 11.0 | 4.9 | 8.1 | 6.0 | 3.6
  Change within +/- 4% | 87.8 | 90.2 | 89.5 | 89.3 | 92.8
  Increase > 4% | 1.2 | 4.9 | 2.3 | 4.8 | 3.6
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.1021, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.428, 95% CI 2-sided [0.155 to 1.184] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.4318, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.682, 95% CI 2-sided [0.262 to 1.773] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0934, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.412, 95% CI 2-sided [0.146 to 1.161] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0317, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.313, 95% CI 2-sided [0.108 to 0.903] — Odds ratio lower than 1 favours the treatment group over placebo

10. Secondary Outcome: Absolute Change From Baseline in PaO2
Description: Absolute change from baseline in Arterial oxygen partial pressure (PaO2) at week 52. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: OC-Randomised set
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 58 | 56 | 64 | 68 | 51
mmHg | -1.69 (1.790) | -2.77 (1.865) | -3.00 (1.686) | -1.46 (1.632) | -0.76 (1.854)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.6443, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-5.66 to 3.51], Standard Error of Mean 2.330 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.5656, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-5.80 to 3.18], Standard Error of Mean 2.280 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.9181, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-4.18 to 4.64], Standard Error of Mean 2.240 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.6970, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-3.77 to 5.63], Standard Error of Mean 2.387 — Mean difference to placebo is calculated. Negative change indicates worsening

11. Secondary Outcome: Absolute Change From Baseline in P(A-a)O2
Description: Absolute change from baseline in Alveolo-arterial oxygen gradient (P(A-a)O2) at week 52. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: OC-Randomised set
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 56 | 54 | 64 | 67 | 51
mmHg | 1.21 (1.898) | 1.27 (1.984) | 2.22 (1.773) | 1.62 (1.723) | 2.56 (1.944)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.9811, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-4.84 to 4.96], Standard Error of Mean 2.490 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6772, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-3.74 to 5.75], Standard Error of Mean 2.412 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.8631, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-4.27 to 5.09], Standard Error of Mean 2.379 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.5942, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-3.62 to 6.31], Standard Error of Mean 2.523 — Mean difference to placebo is calculated. Negative change indicates worsening

12. Secondary Outcome: Absolute Change From Baseline in PaCO2
Description: Absolute change from baseline in Arterial carbon dioxyde partial pressure (PaCO2) at week 52. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: OC-Randomised set
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 58 | 56 | 64 | 68 | 51
mmHg | -0.63 (0.549) | 0.16 (0.573) | -0.44 (0.517) | -0.74 (0.500) | -0.77 (0.569)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.2716, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.62 to 2.19], Standard Error of Mean 0.715 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.7871, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.18 to 1.56], Standard Error of Mean 0.696 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.8721, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-1.46 to 1.24], Standard Error of Mean 0.685 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.8523, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.58 to 1.31], Standard Error of Mean 0.734 — Mean difference to placebo is calculated. Negative change indicates worsening

13. Secondary Outcome: Absolute Change From Baseline in PaO2 by Categories
Description: Absolute change from baseline in Arterial oxygen partial pressure (PaO2) by below mentioned categories:
  1. Decrease > 4 mmHg
  2. Change within +/- 4 mmHg
  3. Increase > 4 mmHg
Time Frame: Baseline and 52 weeks
Population: OC - Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 58 | 56 | 64 | 68 | 51
percentage of participants
  Decrease > 4 mmHg | 34.5 | 50.0 | 42.2 | 39.7 | 29.4
  Change within +/- 4 mmHg | 50.0 | 21.4 | 32.8 | 30.9 | 43.1
  Increase > 4 mmHg | 15.5 | 28.6 | 25.0 | 29.4 | 27.5
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7997, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.093, 95% CI 2-sided [0.549 to 2.175] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.7989, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.916, 95% CI 2-sided [0.467 to 1.797] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.4596, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.780, 95% CI 2-sided [0.403 to 1.508] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.2548, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.665, 95% CI 2-sided [0.330 to 1.341] — Odds ratio lower than 1 favours the treatment group over placebo

14. Secondary Outcome: Absolute Change From Baseline in P(A-a) O2 by Categories
Description: Absolute change from baseline in Alveolo-arterial oxygen gradient (P(A-a) O2) by below mentioned categories:
  1. Decrease > 4 mmHg
  2. Change within +/- 4 mmHg
  3. Increase > 4 mmHg
Time Frame: Baseline and 52 weeks
Population: OC - Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 56 | 54 | 64 | 67 | 51
percentage of participants
  Decrease > 4 mmHg | 25.0 | 37.0 | 31.3 | 25.4 | 17.6
  Change within +/- 4 mmHg | 33.9 | 14.8 | 25.0 | 28.4 | 45.1
  Increase > 4 mmHg | 41.1 | 48.1 | 43.0 | 46.3 | 37.3
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8887, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.051, 95% CI 2-sided [0.521 to 2.122] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.5758, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.216, 95% CI 2-sided [0.613 to 2.410] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.9829, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.993, 95% CI 2-sided [0.506 to 1.949] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.9375, Regression, Logistic; Logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.972, 95% CI 2-sided [0.476 to 1.985] — Odds ratio lower than 1 favours the treatment group over placebo

15. Secondary Outcome: Absolute Change From Baseline in DLCO
Description: Absolute change from Baseline in Diffusing capacity of the lung for carbon monoxide (DLCO) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: mmol.min^-1.kPa^-1
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 75 | 68 | 80 | 81 | 69
mmol.min^-1.kPa^-1 | -0.455 (0.1098) | -0.357 (0.1163) | -0.610 (0.1038) | -0.535 (0.1035) | -0.576 (0.1111)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.4998, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [-0.188 to 0.385], Standard Error of Mean 0.1456 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.2679, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.155, 95% CI 2-sided [-0.430 to 0.120], Standard Error of Mean 0.1399 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.5678, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.080, 95% CI 2-sided [-0.355 to 0.195], Standard Error of Mean 0.1400 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.4053, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.121, 95% CI 2-sided [-0.406 to 0.164], Standard Error of Mean 0.1448 — Mean difference to placebo is calculated. Negative change indicates worsening

16. Secondary Outcome: Absolute Change From Baseline in DLCO by Categories
Description: Absolute change from baseline in Diffusing capacity of the lung for carbon monoxide (DLCO) by below mentioned categories:
  1. Decrease > 15% or > 1
  2. Change <= 15% or <= 1
  3. Increase > 15% or > 1
Time Frame: Baseline and 52 weeks
Population: LOCF Randomized set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 75 | 68 | 80 | 81 | 69
percentage of patients
  Decrease > 15% or > 1 | 37.3 | 38.2 | 43.8 | 35.8 | 50.7
  Change <= 15% or <= 1 | 58.7 | 51.5 | 51.3 | 56.8 | 44.9
  Increase > 15% or > 1 | 4.0 | 10.3 | 5.0 | 7.4 | 4.3
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7307, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.892, 95% CI 2-sided [0.465 to 1.710] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.3869, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.317, 95% CI 2-sided [0.706 to 2.458] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.8237, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.931, 95% CI 2-sided [0.498 to 1.741] — Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.1177, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.676, 95% CI 2-sided [0.878 to 3.202] — Odds ratio lower than 1 favours the treatment group over placebo

17. Secondary Outcome: Absolute Change From Baseline in Distance Walk (6-MWT)
Description: Absolute change from baseline in distance walk (6-MWT) at 52 weeks. The 6-Minutes Walk Test (6-MWT) was conducted according to the American Thoracic Society (ATS) Criteria. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Meter
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 69 | 61 | 75 | 72 | 63
Meter | -35.67 (12.732) | -46.91 (13.652) | -48.84 (11.974) | -36.80 (12.131) | -29.35 (12.957)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.5111, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Median Difference (Final Values) = -11.24, 95% CI 2-sided [-44.86 to 22.37], Standard Error of Mean 17.089 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.4176, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -13.17, 95% CI 2-sided [-45.11 to 18.76], Standard Error of Mean 16.234 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.9454, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-33.60 to 31.34], Standard Error of Mean 16.506 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.7101, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 6.32, 95% CI 2-sided [-27.08 to 39.72], Standard Error of Mean 16.980 — Mean difference to placebo is calculated. Negative change indicates worsening

18. Secondary Outcome: Absolute Change From Baseline in Dyspnoea Rating on Borg Scale Before Exercise (6-MWT)
Description: Absolute change from baseline in Dyspnoea rating before exercise (6-MWT) at 52 weeks based on Borg scale as mentioned below :
  0: Nothing at all, 0.5: Very, very slight (just noticable), 1: Very slight, 2: Slight (light), 3: Moderate, 4: Somewhat severe, 5: Severe (heavy), 6, 7:Very severe, 8, 9, 10: Very, very severe (Maximal).
  The 6-Minutes Walk Test (6-MWT) was conducted according to the ATS Criteria. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 69 | 61 | 75 | 72 | 63
Units on a scale | 0.227 (0.1695) | 0.282 (0.1817) | 0.045 (0.1594) | 0.260 (0.1612) | 0.086 (0.1736)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8090, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.055, 95% CI 2-sided [-0.392 to 0.502], Standard Error of Mean 0.2271 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.3995, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-0.606 to 0.242], Standard Error of Mean 0.2158 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.8822, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.399 to 0.464], Standard Error of Mean 0.2193 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.5338, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.141, 95% CI 2-sided [-0.584 to 0.303], Standard Error of Mean 0.2257 — Mean difference to placebo is calculated. Positive change indicates worsening

19. Secondary Outcome: Change From Baseline in Dyspnoea Rating on Borg Scale After Exercise (6-MWT)
Description: Change from baseline in Dyspnoea rating after exercise (6-MWT) at 52 weeks based on Borg scale as mentioned below :
  0: Nothing at all, 0.5: Very, very slight (just noticable), 1: Very slight, 2: Slight (light), 3: Moderate, 4: Somewhat severe, 5: Severe (heavy), 6, 7:Very severe, 8, 9, 10: Very, very severe (Maximal).
  The 6-Minutes Walk Test (6-MWT) was conducted according to the ATS Criteria. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 69 | 61 | 75 | 72 | 63
Units on a scale | 0.527 (0.2439) | 0.639 (0.2616) | 0.449 (0.2295) | 0.377 (0.2321) | 0.194 (0.2492)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7329, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [-0.532 to 0.755], Standard Error of Mean 0.3272 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.8009, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.078, 95% CI 2-sided [-0.690 to 0.533], Standard Error of Mean 0.3109 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.6358, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.150, 95% CI 2-sided [-0.771 to 0.472], Standard Error of Mean 0.3159 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.3064, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.333, 95% CI 2-sided [-0.973 to 0.307], Standard Error of Mean 0.3252 — Mean difference to placebo is calculated. Positive change indicates worsening

20. Secondary Outcome: Absolute Change From Baseline in MRC Dyspnea Scale by Categories
Description: Absolute change from baseline in Medical Research Council (MRC) dyspnea scale by below mentioned categories:
  1. Decrease
  2. No Change
  3. Increase
Time Frame: Baseline and 52 weeks
Population: LOCF- Randomised
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 77 | 75 | 81 | 82 | 76
percentage of participants
  Decrease | 7.8 | 13.3 | 8.6 | 14.6 | 11.8
  No Change | 51.9 | 45.3 | 53.1 | 45.1 | 53.9
  Increase | 40.3 | 41.3 | 38.3 | 40.2 | 34.2
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.9646, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.014, 95% CI 2-sided [0.540 to 1.906] — Odds ratio lower than 1 favours the treatment group over placebo. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.9850, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 0.994, 95% CI 2-sided [0.536 to 1.844] — Odds ratio lower than 1 favours the treatment group over placebo. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.7136, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.123, 95% CI 2-sided [0.604 to 2.089] — Odds ratio lower than 1 favours the treatment group over placebo. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.1705, Regression, Logistic; An ordinal logistic regression model with fixed terms for treatment, baseline of corresponding continuous value, region; Odds Ratio (OR) = 1.551, 95% CI 2-sided [0.828 to 2.906] — Odds ratio lower than 1 favours the treatment group over placebo. Negative change indicates worsening

21. Secondary Outcome: Absolute Change From Baseline in FEV1/FVC
Description: Change from baseline of percentage of FVC expelled in the first second of a forced expiration (FEV1/FVC) at 52 weeks.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: percentage of FVC
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 84 | 85 | 86 | 85 | 84
percentage of FVC | 1.25 (0.529) | -0.10 (0.533) | 0.00 (0.511) | -0.53 (0.516) | -0.42 (0.513)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.0479, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-2.69 to -0.01], Standard Error of Mean 0.680 — Mean difference to placebo is calculated
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.0685, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-2.58 to 0.09], Standard Error of Mean 0.680 — Mean difference to placebo is calculated
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0099, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-3.12 to -0.43], Standard Error of Mean 0.684 — Mean difference to placebo is calculated
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0152, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -1.67, 95% CI 2-sided [-3.01 to -0.32], Standard Error of Mean 0.683 — Mean difference to placebo is calculated

22. Secondary Outcome: Change From Baseline in SGRQ Total Score
Description: Change from baseline in Saint George's Respiratory Questionnaire (SGRQ) total score. Total score is defined as sum of the three domain scores symptoms, activities and impacts. Scores range from 0 to 100, with higher scores indicating worst possible health status.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 79 | 76 | 82 | 82 | 75
units on a scale | 5.46 (1.731) | 4.67 (1.779) | 2.18 (1.654) | 1.48 (1.660) | -0.66 (1.712)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7250, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-5.22 to 3.64], Standard Error of Mean 2.253 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.1389, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -3.28, 95% CI 2-sided [-7.63 to 1.07], Standard Error of Mean 2.213 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0741, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -3.98, 95% CI 2-sided [-8.35 to 0.39], Standard Error of Mean 2.221 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0071, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -6.12, 95% CI 2-sided [-10.57 to -1.67], Standard Error of Mean 2.262 — Mean difference to placebo is calculated. Positive change indicates worsening

23. Secondary Outcome: Change From Baseline in SGRQ Domain Score Symptoms
Description: Change from baseline in Saint George's Respiratory Questionnaire (SGRQ) domain score symptoms. Scores range from 0 to 100, with higher scores indicating more limitations.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 79 | 76 | 82 | 82 | 76
units on a scale | 6.45 (2.446) | 3.39 (2.514) | 2.11 (2.338) | 2.33 (2.346) | -3.14 (2.403)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.3370, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -3.06, 95% CI 2-sided [-9.32 to 3.20], Standard Error of Mean 3.183 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.1659, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -4.34, 95% CI 2-sided [-10.49 to 1.81], Standard Error of Mean 3.126 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1897, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -4.12, 95% CI 2-sided [-10.29 to 2.05], Standard Error of Mean 3.138 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0028, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -9.60, 95% CI 2-sided [-15.86 to -3.34], Standard Error of Mean 3.184 — Mean difference to placebo is calculated. Positive change indicates worsening

24. Secondary Outcome: Change From Baseline in SGRQ Domain Score Impacts
Description: Change from baseline in Saint George's Respiratory Questionnaire (SGRQ) domain score impacts. Scores range from 0 to 100, with higher scores indicating worst possible health status.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF - Randomised set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 79 | 76 | 82 | 82 | 75
units on a scale | 4.21 (1.986) | 3.71 (2.040) | 1.73 (1.897) | 0.79 (1.906) | -0.14 (1.965)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8458, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-5.59 to 4.58], Standard Error of Mean 2.586 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.3286, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-7.48 to 2.51], Standard Error of Mean 2.540 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1799, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -3.42, 95% CI 2-sided [-8.43 to 1.59], Standard Error of Mean 2.548 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0948, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -4.35, 95% CI 2-sided [-9.46 to 0.76], Standard Error of Mean 2.597 — Mean difference to placebo is calculated. Positive change indicates worsening

25. Secondary Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Domain Score Activities
Description: Change from baseline in Saint George's Respiratory Questionnaire (SGRQ) domain score activities. Scores range from 0 to 100, with higher scores indicating worst possible health status.
  Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 79 | 76 | 82 | 82 | 75
units on a scale | 7.48 (1.910) | 7.39 (1.962) | 3.54 (1.824) | 3.00 (1.832) | 0.32 (1.887)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.9708, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-4.98 to 4.79], Standard Error of Mean 2.484 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.1069, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-8.74 to 0.85], Standard Error of Mean 2.440 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0682, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -4.49, 95% CI 2-sided [-9.31 to 0.34], Standard Error of Mean 2.453 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0043, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -7.16, 95% CI 2-sided [-12.06 to -2.26], Standard Error of Mean 2.494 — Mean difference to placebo is calculated. Positive change indicates worsening

26. Secondary Outcome: St George's Respiratory Questionnaire (SGRQ) Responder
Description: St George's Respiratory Questionnaire (SGRQ) responder (<= -4 points change) (%) at 52 weeks-worst case
Time Frame: 52 weeks
Population: Worst case - Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
percentage of participants | 16.1 | 23.0 | 26.7 | 32.6 | 29.1
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.2698, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel test to adjust for region effect; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.72 to 3.31] — In case of missing data, patient has been set to non-responder. Odds ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.0891, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel test to adjust for region effect; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.90 to 4.01] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0069, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel test to adjust for region effect; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.29 to 5.66] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0341, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel test to adjust for region effect; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.05 to 4.61] — [estimate comment as in outcome 26, analysis 1]

27. Secondary Outcome: Change From Baseline in TLC
Description: Change from Baseline in Total Lung Capacity (TLC) at 52 weeks. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 75 | 68 | 80 | 80 | 69
Liters | -0.240 (0.0765) | -0.218 (0.0809) | -0.100 (0.0725) | -0.082 (0.0723) | 0.118 (0.0774)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8288, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.178 to 0.222], Standard Error of Mean 0.1015 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.1506, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [-0.051 to 0.332], Standard Error of Mean 0.0974 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1059, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.158, 95% CI 2-sided [-0.034 to 0.351], Standard Error of Mean 0.0977 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.358, 95% CI 2-sided [0.160 to 0.556], Standard Error of Mean 0.1008 — Mean difference to placebo is calculated. Negative change indicates worsening

28. Secondary Outcome: Change From Baseline in RV
Description: Change from Baseline in Residual volume (RV) at 52 weeks. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 75 | 68 | 80 | 80 | 69
Liters | -0.036 (0.0512) | -0.056 (0.0543) | 0.029 (0.0484) | -0.012 (0.0484) | 0.086 (0.0518)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7789, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.153 to 0.115], Standard Error of Mean 0.0680 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.3149, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.063 to 0.194], Standard Error of Mean 0.0652 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.7062, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.025, 95% CI 2-sided [-0.104 to 0.153], Standard Error of Mean 0.0654 — Mean difference to placebo is calculated. Positive change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0703, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.123, 95% CI 2-sided [-0.010 to 0.255], Standard Error of Mean 0.0675 — Mean difference to placebo is calculated. Positive change indicates worsening

29. Secondary Outcome: Change From Baseline in TGV
Description: Change from Baseline in Thoracic gas volume (TGV) at 52 weeks. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 73 | 64 | 78 | 78 | 66
Liters | -0.137 (0.0657) | -0.075 (0.0707) | -0.035 (0.0622) | -0.016 (0.0623) | 0.200 (0.0668)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.4792, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [-0.111 to 0.236], Standard Error of Mean 0.0884 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.2221, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.103, 95% CI 2-sided [-0.062 to 0.268], Standard Error of Mean 0.0839 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1510, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [-0.044 to 0.287], Standard Error of Mean 0.0843 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0001, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.337, 95% CI 2-sided [0.165 to 0.509], Standard Error of Mean 0.0874 — Mean difference to placebo is calculated. Negative change indicates worsening

30. Secondary Outcome: Change From Baseline in VC
Description: Change from baseline in Vital capacity (VC) at 52 weeks. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 74 | 67 | 80 | 80 | 69
Liters | -0.191 (0.0458) | -0.095 (0.0485) | -0.107 (0.0433) | -0.082 (0.0432) | 0.010 (0.0462)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.1129, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [-0.023 to 0.217], Standard Error of Mean 0.0609 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.1498, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.084, 95% CI 2-sided [-0.031 to 0.199], Standard Error of Mean 0.0584 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0632, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.109, 95% CI 2-sided [-0.006 to 0.224], Standard Error of Mean 0.0585 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0009, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.201, 95% CI 2-sided [0.083 to 0.320], Standard Error of Mean 0.0604 — Mean difference to placebo is calculated. Negative change indicates worsening

31. Secondary Outcome: Change From Baseline in IC
Description: Change from Baseline in Inspiratory Capacity (IC) at 52 weeks. Means were adjusted based on an ANCOVA with fixed terms for treatment, baseline, region.
Time Frame: Baseline and 52 weeks
Population: LOCF-Randomised set
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 74 | 67 | 78 | 80 | 68
Liters | -0.031 (0.0509) | -0.064 (0.0539) | -0.053 (0.0483) | -0.038 (0.0479) | -0.012 (0.0515)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.6306, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.033, 95% CI 2-sided [-0.165 to 0.100], Standard Error of Mean 0.0676 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.7426, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.021, 95% CI 2-sided [-0.149 to 0.106], Standard Error of Mean 0.0650 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.9209, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.134 to 0.121], Standard Error of Mean 0.0651 — Mean difference to placebo is calculated. Negative change indicates worsening
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.7701, ANCOVA; ANCOVA with fixed terms for treatment, baseline, region; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.112 to 0.152], Standard Error of Mean 0.0671 — Mean difference to placebo is calculated. Negative change indicates worsening

32. Secondary Outcome: Number of Patients With at Least One IPF Exacerbation
Description: Number of patients with at least one Idiopathic Pulmonary Fibrosis (IPF) exacerbation at 52 weeks
Time Frame: 52 weeks
Population: OC-Randomised set
Measure: Number; unit: participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
participants | 12 | 10 | 10 | 6 | 2
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.6671, Negative binomial model — Based on the statistic of ln(risk ratio) having a normal distribution N[0,[ (1/number with at least one exacerbation in Nintedanib group) + (1//number with at least one exacerbation in placebo) ] ]; Default log link function and adjusted for an off-set variable (logarithm of the follow-up time), for gender, height, age and region as fixed effects; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.36 to 1.93] — Risk ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.5926, Negative binomial model — [p-value comment as in outcome 32, analysis 1]; [statistical method as in outcome 32, analysis 1]; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.34 to 1.84] — Risk ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1381, Negative binomial model — [p-value comment as in outcome 32, analysis 1]; [statistical method as in outcome 32, analysis 1]; Risk Ratio (RR) = 0.48, 95% CI 2-sided [0.18 to 1.27] — Risk ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0150, Negative binomial model — [p-value comment as in outcome 32, analysis 1]; [statistical method as in outcome 32, analysis 1]; Risk Ratio (RR) = 0.16, 95% CI 2-sided [0.03 to 0.70] — Risk ratio lower than 1 favours the treatment group over placebo

33. Secondary Outcome: Occurrences of IPF Exacerbations Per Patient Per Year
Description: Occurrences of Idiopathic Pulmonary Fibrosis (IPF) exacerbations per patient per year at 52 weeks
Time Frame: 52 weeks
Population: OC-Randomised set
Measure: Mean (Standard Deviation); unit: Exacerbations Per Year
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
Exacerbations Per Year | 0.243 (0.8008) | 0.243 (0.7884) | 0.242 (0.9830) | 0.256 (1.7315) | 0.075 (0.5177)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.8282, Negative binomial model; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.347 to 2.336] — Risk ratio is actually Rate Ratio. Rate ratio is calculated based on Negative binomial model with default log link function and adjusted for an off-set variable and age, height, gender, region (all effects fixed)
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.5326, Negative Binomial model; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.278 to 1.938] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1944, Negative Binomial model; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.167 to 1.438] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0324, Negative Binomial model; Risk Ratio (RR) = 0.22, 95% CI 2-sided [0.056 to 0.882] — [estimate comment as in outcome 33, analysis 1]

34. Secondary Outcome: Time to First Occurrence of IPF Exacerbation
Description: This endpoint is called time to first occurrence of IPF exacerbation however it was actually analysed as the proportion of patients having occurrence of Idiopathic Pulmonary Fibrosis (IPF) exacerbation at 52 weeks.
  Failure means participants with event and Censored means participants with no event.
Time Frame: 52 weeks
Population: OC-Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
percentage of participants
  Failure | 13.8 | 11.5 | 11.6 | 7.0 | 2.3
  Censored | 86.2 | 88.5 | 88.4 | 93.0 | 97.7
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.5206, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.758, 95% CI 2-sided [0.326 to 1.765] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.6862, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.841, 95% CI 2-sided [0.362 to 1.952] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.1891, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.517, 95% CI 2-sided [0.193 to 1.384] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0161, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.158, 95% CI 2-sided [0.035 to 0.711] — Hazard ratio lower than 1 favours the treatment group over placebo

35. Secondary Outcome: Survival (Death Due to Respiratory Cause, and Lung-transplant Free)
Description: Survival (death due to respiratory cause, and lung-transplant free) at 52 weeks.
  Failure means participants with event and Censored means participants with no event.
Time Frame: 52 weeks
Population: OC-Randomised set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
percentage of participants
  Failure | 9.2 | 10.3 | 3.5 | 2.3 | 2.3
  Censored | 90.8 | 89.7 | 96.5 | 97.7 | 97.7
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7449, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 1.173, 95% CI 2-sided [0.448 to 3.072] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.0925, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.316, 95% CI 2-sided [0.083 to 1.209] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.0379, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.190, 95% CI 2-sided [0.040 to 0.911] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.0600, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.225, 95% CI 2-sided [0.048 to 1.065] — Hazard ratio lower than 1 favours the treatment group over placebo

36. Secondary Outcome: Time to Progression
Description: Time to progression. Progression was defined as at least one of the following: 5mmHg increase in the alveolo-arterial pressure difference in oxygen (P(A-a)O2), 10% decrease in FVC (FVC(baseline)-FVC(progression) >= 10%) or Death.
  Failure means participants with event and Censored means participants with no event.
Time Frame: 52 weeks
Population: OC - Randomised set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86
Days | 363 [302 to 366] | 365 [309 to 366] | 365 [330 to 365] | 365 [NA to NA] — The 95% CI for the median could not be calculated due to computational reason as the number of participants with event was insufficient. | 365 [NA to NA] — The 95% CI for the median could not be calculated due to computational reason as the number of participants with event was insufficient.
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 50 qd; Test type: Superiority or Other; p = 0.7883, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 1.055, 95% CI 2-sided [0.713 to 1.563] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 2: Comparison: Placebo vs Nintedanib 50 Bid; Test type: Superiority or Other; p = 0.8293, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.958, 95% CI 2-sided [0.646 to 1.419] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 3: Comparison: Placebo vs Nintedanib 100 Bid; Test type: Superiority or Other; p = 0.3030, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.805, 95% CI 2-sided [0.534 to 1.216] — Hazard ratio lower than 1 favours the treatment group over placebo
Statistical Analysis 4: Comparison: Placebo vs Nintedanib 150 Bid; Test type: Superiority or Other; p = 0.6505, Regression, Cox; Cox regression model with fixed terms for treatment, gender, age, height, region; Hazard Ratio (HR) = 0.910, 95% CI 2-sided [0.605 to 1.369] — Hazard ratio lower than 1 favours the treatment group over placebo

37. Secondary Outcome: Pre-dose Plasma Concentration of Nintedanib in Plasma at Steady State on Day 365 (Cpre,ss,365) and Day 729 (Cpre,ss,729).
Description: Cpre,ss,729 represents the pre-dose plasma concentration of nintedanib in plasma at steady state on Day 729 and Cpre,ss,365 represents the pre-dose plasma concentration of nintedanib in plasma at steady state on Day 365. At day 365, values only for Nintedanib 50 qd group are presented as no values reported for other groups and at day 729, values are presented for all group except for Nintedanib 50 qd group as no values reported for it.
Time Frame: day 365 and day 729
Population: Randomised set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Number analyzed (Participants) | 35 | 52 | 53 | 33
ng/mL | 1.07 (41.6) | 2.12 (91.1) | 4.20 (69.0) | 6.66 (94.0)

ADVERSE EVENTS:
Time Frame: First drug administration until 14 days after last drug administration
Arm/Group | Placebo | Nintedanib 50 qd | Nintedanib 50 Bid | Nintedanib 100 Bid | Nintedanib 150 Bid
Serious Adverse Events (participants affected / at risk) | 26/85 | 26/86 | 23/86 | 18/86 | 23/85
Other Adverse Events (participants affected / at risk) | 51/85 | 52/86 | 55/86 | 64/86 | 57/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | Nintedanib 50 qd (N=86) | Nintedanib 50 Bid (N=86) | Nintedanib 100 Bid (N=86) | Nintedanib 150 Bid (N=85)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 2 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Scleritis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 2 | 1 | 1
Campylobacter intestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 2 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 1 | 2 | 2 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
PO2 decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Pulmonary arterial pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Transplant evaluation (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephritic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 6 | 4 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Lung transplant (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Prosthesis implantation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | Nintedanib 50 qd (N=86) | Nintedanib 50 Bid (N=86) | Nintedanib 100 Bid (N=86) | Nintedanib 150 Bid (N=85)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 3 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 5 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6 | 10 | 2 | 10
Diarrhoea (Gastrointestinal disorders) | 13 | 8 | 16 | 32 | 44
Nausea (Gastrointestinal disorders) | 8 | 9 | 7 | 17 | 20
Vomiting (Gastrointestinal disorders) | 4 | 1 | 4 | 11 | 11
Fatigue (General disorders) | 7 | 4 | 5 | 8 | 9
Bronchitis (Infections and infestations) | 9 | 10 | 14 | 6 | 8
Influenza (Infections and infestations) | 4 | 1 | 3 | 1 | 6
Lower respiratory tract infection (Infections and infestations) | 6 | 1 | 4 | 6 | 6
Nasopharyngitis (Infections and infestations) | 11 | 11 | 8 | 15 | 6
Sinusitis (Infections and infestations) | 1 | 1 | 7 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 7 | 10 | 12 | 7
Urinary tract infection (Infections and infestations) | 3 | 1 | 4 | 5 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2 | 6
Weight decreased (Investigations) | 0 | 3 | 1 | 3 | 8
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 4 | 4 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 2 | 3 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 5 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 6 | 7 | 6
Headache (Nervous system disorders) | 5 | 7 | 9 | 8 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 17 | 20 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 11 | 11 | 5
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 5 | 5 | 2

LIMITATIONS AND CAVEATS:
There were numerous additional pre-specified endpoints. Full results are available under the BI Transparency web page ( http://trials.boehringer-ingelheim.com/trial_results.html )

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights